CLINICAL TRIAL: NCT06926023
Title: A Prospective, Randomized, Evaluator-blind, Clinical Trial Evaluating the 1550nm Non-ablative Fractional or 1927nm Thulium Fractional Laser for the Treatment of Female Pattern Hair Loss
Brief Title: 1550nm Non-ablative Fractional Vs 1927nm Thulium Fractional Laser for the Treatment of Female Pattern Hair Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hair-1550-vs-1927
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Evaluator Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- GROUP A 1550nm non-ablative fractional laser (Experimental): Group A: Study subjects will have a total of 4 treatments spaced 4 weeks apart. No additional topical treatments applied
  Interventions: Device: 1550nm non-ablative fractional laser
- GROUP B 1927 thulium fractional laser (Active Comparator): Group B: Study subjects will have a total of 4 treatments spaced 4 weeks apart. No additional topical treatments applied.
  Interventions: Device: 1927 thulium fractional laser

INTERVENTIONS:
Device: 1550nm non-ablative fractional laser — Treatment with the 1550nm non-ablative fractional laser for female pattern hair loss to the frontal and crown of scalp.
  Arms: GROUP A 1550nm non-ablative fractional laser
Device: 1927 thulium fractional laser — Treatment with the 1927 thulium fractional laser for female pattern hair loss to the frontal and crown of scalp.
  Arms: GROUP B 1927 thulium fractional laser

SUMMARY:
To evaluate the efficacy of either a 1550nm non-ablative fractional laser or a 1927nm thulium fractional laser in the treatment of female pattern hair loss (FPHL).

DETAILED DESCRIPTION:
The study will have a total of eight visits, from baseline (Day 0) to the final follow-up at 3 months following the last treatment. The first visit (Visit 1, Day 0) will be for screening. During this visit, informed consent, HIPAA authorization, and a photo release will be obtained from all participants. Investigators will review the inclusion and exclusion criteria, medical history, and any concurrent medications. A urine pregnancy test will be administered for all eligible subjects. Baseline hair loss will be evaluated and standardized 2D photographs will be taken for future comparison. Hair count, hair density, and terminal hair average diameter will be evaluated as a pre-defined scalp location.. Patients will be randomized to groups (Group A or B).Visits 2 through 5 (Day 30, 60, 90, and 120, ± 5 days) will consist of the treatment phase. Participants will be treated based on which treatment group they were randomized too as below

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 35-65 years
2. Fitzpatrick skin types I-IV
3. Presence of female pattern hair loss of the frontal or vertex of scalp (Sinclair (II-IV)
4. Must be willing and can comply with all study protocols, including all treatment schedules, follow up visit, assessments, sign a photography release and ICF, and complete the entire course of the study
5. Patients with gray hair roots must be willing to dye their gray hair within two weeks of the first appointment and the last 3-month follow-up visit to ensure consistency in evaluator assessments.
6. No use of hair growth treatments or procedures within 6 months prior to enrollment (including hair supplements such as Nutrafol)
7. Subjects in good general health based on investigator's judgment and medical history
8. Negative urine pregnancy test result at the time of study entry
9. Subjects will be of non-childbearing potential defined as:
10. Having no uterus
11. No menses for at least 12 months.
12. Or;
13. Subjects of childbearing potential must agree to use an effective method of birth control during the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation. Acceptable forms of birth control below:
14. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
15. Intrauterine coil
16. Bilateral tubal ligation
17. Hysterectomy
18. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
19. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
20. Vasectomized (must agree to use barrier method described above (4) if becomes sexually active with un-vasectomized partner).

Exclusion Criteria:

1. No surgery, pregnancy, breast feeding, change in or addition of hormonal contraception in the last 6 months
2. No history of iron deficiency anemia, vitamin D deficiency, or thyroid disease (hypothyroidism or hyperthyroidism or currently on thyroid supplementation)
3. Use of scalp light or with laser treatment within the last 6 months.
4. Use of topical or systemic drugs affecting hair growth within 6 months prior to enrollment (such as oral spironolactone, finasteride, oral or topical minoxidil, and supplements marketed for hair growth such as Nutrafol)
5. Supplementation of oral tumeric/curcumin
6. History of hair transplant
7. Systemic or scalp disease that may affect hair growth (Lupus, alopecia areata, folliculitis decalvans, psoriasis, scalp infection, seborrheic dermatitis, CCCA, telogen effluvium)
8. Pregnancy or planned pregnancy during the study or currently breastfeeding.
9. Any uncontrolled systemic disease
10. History of autoimmune connective tissue disease or thyroid disease.
11. Current use of immunosuppressive medication.
12. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
13. Active dermatitis, metal or other active implants, active infection in the proposed treatment area.
14. Subjects with scarring in the treatment areas (scalp) Subjects with a history of keloids will be excluded.
15. History of bleeding disorder, concomitant use of anticoagulants, history of connective tissue disease, history of Bell's Palsy, epilepsy, smoking, pregnancy, and lactation.
16. Inability to following the comply with study protocols and regulations
17. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Identity
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in hair count at a predefined 1cm x 1cm scalp location | Baseline and Day 180
  Measured by the Canfield Hair Matrix System
Change in hair density (hairs/cm) at the same predefined scalp area | Baseline and Day 180
  Measured by the Canfield Hair Matrix System
Change in terminal hair average diameter (in mm) at the predefined location | Baseline and Day 180
  Measured by the Canfield Hair Matrix System

SECONDARY OUTCOMES:
Change in Sinclair Scale score | Baseline and Day 180
  Sinclair photo grading scale II-IV Grades 1 thru 5 (system would not allow to paste/insert the photo scale)
Change in perceived age based on blinded evaluator assessment of global scalp photographs | Baseline and Day 180
  Estimated age based on posterior scalp evaluation
  Visit Perceived Age (years)
Subjective Assessment on Hair outcomes | Day 180
  Category 1 - No improvement 2 - Slight improvement 3 - Moderate improvement 4 - Noticeable improvement 5 - Significant improvement
  Hair Density
  Hair Thickness
  Hair Growth
Physician Global Aesthetic Improvement Scale (PGAIS) via photos by blinded evaluator | Day 180
  Description Grade Much Improved 2 Improved 1 No Change 0 Worse -1 Much Worse -2
Comfort Level Visual Analog Scale | Baseline, Day 30, Day 60, Day 90
  0 No Pain 1-3 Mild 4-6 Moderate to Severe 7-9 Very Severe 10 Worst Pain Possible

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center/Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided